CLINICAL TRIAL: NCT04444258
Title: Development and Use of Virtual Reality Application in Teaching Fetal Development
Brief Title: Teaching Fetal Development With Virtual Reality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Reyhan Aydin Doğan, Prelector, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2020/263
Record Dates: First submitted 2020-06-18; First posted 2020-06-23 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Educational Problems
Keywords: virtual reality; midwifery student education; virtual pregnancy

STUDY DESIGN:
Intervention Model Description: The sample will consist of 105 midwifery students, including 35 control, 35 experiment I and 35 experiment II, as a result of the G-power analysis calculated by 0.95 power, among the midwifery students who took theoretical 4 hours in their curriculum within the scope of the week of week, including fetal development.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental I Group (Experimental): After the Fetal Development Assessment Information Form (FEGBF), a computer-aided and guided virtual reality application prepared by the researchers including the phases of the fetus week by week will be watched and then FEGBF will be applied again by changing the locations of the questions.
  Interventions: Other: Application of computer aided virtual reality glasses; Other: Teaching fetal development theoretically
- Control Group (No Intervention): FEGBF will be applied after 4 hours of theory training. Virtual pregnancy application will not be watched.

INTERVENTIONS:
Other: Application of computer aided virtual reality glasses — Experimental I Group: After the Fetal Development Assessment Information Form (FEGBF), a computer-aided and guided virtual reality application prepared by the researchers including the phases of the fetus week by week will be watched and then FEGBF will be applied again by changing the locations of the questions.
  Arms: Experimental I Group
Other: Teaching fetal development theoretically — Control Group: FEGBF will be applied after 4 hours of theory training. Virtual pregnancy application will not be watched.
  Arms: Experimental I Group

SUMMARY:
In this study, it was aimed to design virtual pregnancy for pregnancy formation, fetal and placental development in the virtual reality environment and to evaluate the effectiveness of the designed virtual pregnancy on midwifery education.

Our study, which will be the first in our second country in the world, aims to reduce the application errors and determine deviations from normal by examining the formation of pregnancy, maternal, fetal and placental changes, which form the basis of midwifery profession, before having clinical experience. In this direction, the objectives of our study are;

* Development of the virtual pregnancy application, which will be designed for the first time in our country,
* Ensuring the effective use of virtual pregnancy practice in midwifery education,
* Visualizing fetal and placental development with virtual pregnancy that will form the basis of midwifery education,
* To minimize the application errors experienced in clinical practices of midwifery students,
* To increase educational effectiveness, clinical and academic success by visualizing the formation of pregnancy.
* Measuring cognitive loadings of students after education
* Measuring students' sense of readiness

DETAILED DESCRIPTION:
Today, simulation education is gradually increasing and it is used effectively in the field of midwifery education (1). It is observed that simulation education is used effectively during midwifery, pregnancy, delivery or postpartum period (2,9). Providing a virtual reality perspective to midwifery simulation training will enable students to use midwifery practices effectively before going to clinical practice (3,5). Teaching of pregnancy, which forms the basis of midwifery education, with virtual reality application will minimize clinical application errors and will provide early diagnosis of fetal presentation and placental anomalies that will be able to experience pregnancy and childbirth. They will be able to effectively see the differences that occur as pregnancy progresses and the maternal-fetal response to these differences. It is an up-to-date and important subject that will enable them to see the pregnancy process, maternal-fetal development, placental differences and mother's circulatory response in three dimensions without any obstacle in midwifery education with virtual pregnancy application (4,6,7,8,9).

Since this application is a newly developed technique, it will create a current perspective on midwifery education and fill the gap in the virtual reality simulation in its education, and will provide a basis for midwifery education and literature. Although there are studies on simulation in midwifery or health in our country, there is no study that combines and applies virtual reality and pregnancy in midwifery. In the studies related to virtual reality and health field and midwifery profession in the world, the profession of virtual reality has been supported in studies that have positive effects on education.

Type of the Study: The study is planned to be an experimental study designed as an experimental and control group.

Location and Date of the Research: The study will be conducted in the Midwifery Department of the Faculty of Health Sciences of Karabuk University and between November 2019 and October 2020.

The research consists of 2 parts. In Part I, Virtual Reality Application will be Developed. Virtual pregnancy software will be prepared through service procurement. For this, fetal development and fetal physiology will be written in detail by researchers week by week and virtual pregnancy will be created.

II. The application of the research will be done in the department.

SECTION I: Development of Virtual Reality Application

In the 1st part of the research, the software of virtual pregnancy will be prepared through service procurement. For this, algorithms will be created by researchers in detail by writing fetal development, fetal physiology and anatomy weekly. This algorithm will be transferred to the glasses based on images and drawings (10,11) of fetal development weekly and weekly images of fetal development from the book of Obstetrics and Gynecology, and the images shared on the internet for fetal development. As stated in the budget form, service will be purchased for the development of the Virtual Pregnancy software. TUBITAK will be applied for this service.

With the Virtual Pregnancy application,

* Learning pregnancy formation week by week,
* To follow placental development and to understand deviations from normal,
* It will provide the opportunity to learn normal fetal development and besides, information will be remembered for a long time. In this way, its effectiveness in virtual pregnancy midwifery education will be evaluated.

II. Department: Application of the Research

In this last part of the research, the application part of the research has been started. The research will consist of 3 groups, 2 experimental groups and a control group. 35 students will be admitted to each group as a result of G-power analysis calculated with 0.95 power.

The Universe of the research will consist of 464 Midwifery students studying at Karabuk University.

The sample will consist of 105 midwifery students, including 35 control, 35 experiment I and 35 experiment II, as a result of the G-power analysis calculated by 0.95 power, among the midwifery students who took theoretical 4 hours in their curriculum within the scope of the week of week, including fetal development.

Experimental I Group: After the Fetal Development Assessment Information Form (FEGBF), a computer-aided and guided virtual reality application prepared by the researchers including the phases of the fetus week by week will be watched and then FEGBF will be applied again by changing the locations of the questions.

Experiment II Group: Following the Fetal Development Assessment Information Form (FEGBF), the computer-aided and unguided virtual reality application prepared by the researchers including the fetal development week by week will be monitored, and then FEGBF will be applied again by changing the locations of the questions.

Control Group: FEGBF will be applied after 4 hours of theory training. Virtual pregnancy application will not be watched.

At the first stage: after 4 hours of theory training to all three groups, the information form (FEGBF) prepared by the researchers to be used in this research will be applied as the first test.

In the second stage: No application will be made to the control group, computer-aided and guided virtual reality application will be applied to the experimental group, and computer-free and non-guided virtual application will be monitored to the experiment II group.

In the third phase: Post-tests will be applied by changing the locations of FEGBF questions. After the 4-hour theory training for the control group, the posttest will be done after the virtual birth application is watched on the experiment groups. Also, at this stage, "Cognitive Load Scale" and "Feel of Inventory" will be applied to the experimental groups after the application.

In the fourth stage: After 6 weeks, all three groups will be relocated to FEGBF, and the effectiveness of the application of virtual birth will be examined in remembering and recalling the information.

In order not to affect the groups determined by the computer-aided randomization program according to the class list order as the experiment and control groups, the students will not be informed which one is in the experiment and which is in the control group. Since virtual pregnancy application will be applied to all experimental group students on the same day, the possibility of students being affected by each other will be excluded.

Students who could not participate in the study and were selected as a control group in randomization will also be provided with virtual reality glasses after the study, so that all students will see the virtual birth application and equality will be achieved.

Randomization of the Study: The class list of the students who agree to participate in the study will be transferred to the computer supported randomization program and the groups will be determined. Sufficient sample size will be provided by choosing again from the students who did not participate in the study for the last minute or who did not participate in the study for reasons such as disease or control group, who accepted to participate in the study and were not selected in randomization.

Teaching complex procedural information by simulation may cause cognitive load in learners (6). The way to reduce cognitive load and increase teaching achievements is to establish a sample based system. Thus, the use of rules and examples through modeling simplifies the process of learning complex procedures. For this reason, the directive on the use of VR and sample application videos will be presented to the learners as modeling.

Data Collection Tools:

Data collection form: It is planned to apply a form consisting of 15 questions, which includes the characteristics of the participants such as age, marital status, educational status and family type.

Fetal Development Assessment Information Form (FEGBF): For the preparation of the information form, the latest literature information, midwifery core curriculum (EUÇEP) created by YÖK was reviewed and an information form consisting of 42 questions related to fetal physiology issues and phases of fetal development was prepared. The items in the information form will be presented to the students in the form of a full sentence that can be true or false, and students will be asked to answer these statements as "True" or "False". Total response time is 30 minutes. Correct answers will be evaluated as 1 point, Wrong answers will be evaluated as 0 points. Wrong expressions were also used in the information form, and these items were coded in reverse compared to others. The lowest score to be taken from the information form is 0 and the highest total score is 42.

Cognitive Load Scale: Kılıç et al. (2004) "Cognitive Load Scale" (BYÖ) adapted to Turkish will be used. It has single factor and nine points (very little, very little, little, partly little, neither more nor less, more, more, more, more, more, more or more). The Cronbach Alpha internal consistency coefficient of the original version was found to be 0.90. Kılıç et al. (2004) in the adaptation study, the Cronbach Alpha internal consistency coefficient was found as .78. The lowest point of the scores obtained from the scale is 1.00, the middle point is 5.00 and the highest point is 9.00. Participants scoring below five points were evaluated as "cognitively overloaded", and participants scoring above 5 points were evaluated as "cognitively overloaded" (12).

Availability Sensitivity Scale: It is a scale that was originally 7-likert type in Turkish validity reliability in 2018, but reduced to 5-likert type in Turkish validity. Cronbach Alpha reliability coefficient of the scale was calculated as 0.91. The scale measures the sense of presence in virtual reality-based learning environments. The scale has 5 factors (lower size): Participation (Factor 1), Cohesion / Surrounding (Factor 2), Sensory Commitment (Factor 3), Interaction (Factor 4) and Interface Quality (Factor 5) and consists of 29 questions (13 ).

Ethical Aspect of the Research: The study will start after obtaining the ethics committee permission from the non-interventional research ethics committee of Karabük University, and the informed volunteer consent form will be obtained from each student who agrees to participate in the study.

Data Analysis of the Research: Analysis of the data of the study will be done using IBM SPSS for Mac book 24 version. Average values will be taken for socio-demographic characteristics. In study models with experiment / control groups, the experimental group is tested / tested and finally tested. The same test will be applied to the control group without experiment. Whether the difference between the measurements of the three groups is meaningful or not will be calculated using "z or t test for independent groups". For statistical significance, p <0.05 level will be accepted. While evaluating the study data, frequency distributions for categorical variables and descriptive statistics (mean, standard deviation, median, minimum, maximum) for numerical variables will be used. Whether there is a relationship between two categorical variables will be checked by Chi-Square analysis and whether there is a relationship between two numerical variables will be examined by Pearson Correlation analysis. If the number of groups is two, whether there is a difference between the variables and the scores, it will be tested with the "significance test of the difference between the two averages" (independent t test), and if the group number is more than two, "one way variance analysis" (ANOVA). As a result of the analysis, first of all, the Levene test for variance homogeneity will be checked by the "multiple comparison test" (Bonferroni or Tamhane's T2), from which group or groups the difference originated.

ELIGIBILITY:
Inclusion Criteria:

* Being at least a 4nd year student at the Midwifery Department of
* I. Karabuk University,
* II. 84 midwifery students will be volunteering to participate in the research.

Exclusion Criteria:

* In our study, there are no exclusion criteria.

Min Age: 24 Months | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
To provide midwifery students to learn fetal development week by week | Within 6 weeks after the fetal development virtual reality application is developed and applied.
  All three groups will be developed by researchers after 4 hours of theoretical training; "Fetal Development Assessment Information Form (FEGBF)" will be applied to evaluate fetal development and fetal physiology knowledge.

OTHER OUTCOMES:
Ensuring that virtual reality application in the teaching of Fetal Development focuses students' attention and mental potential on related stimuli, activities or events | Within 6 weeks after the fetal development virtual reality application is developed and applied.
  At this stage, "Cognitive Load Scale" and "Feel of Inventory" will be applied to the experimental groups after the application.

CONTACTS AND LOCATIONS:
Locations (1):
- Karabuk University, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I'm undecided now. I want to decide in the future

REFERENCES:
- [Background] Fealy S, Jones D, Hutton A, Graham K, McNeill L, Sweet L, Hazelton M. The integration of immersive virtual reality in tertiary nursing and midwifery education: A scoping review. Nurse Educ Today. 2019 Aug;79:14-19. doi: 10.1016/j.nedt.2019.05.002. Epub 2019 May 4. PMID 31078869
- [Result] Williams J, Jones D, Walker R. Consideration of using virtual reality for teaching neonatal resuscitation to midwifery students. Nurse Educ Pract. 2018 Jul;31:126-129. doi: 10.1016/j.nepr.2018.05.016. Epub 2018 May 28. PMID 29879636
- [Result] Cooper S, Cant R, Porter J, Bogossian F, McKenna L, Brady S, Fox-Young S. Simulation based learning in midwifery education: a systematic review. Women Birth. 2012 Jun;25(2):64-78. doi: 10.1016/j.wombi.2011.03.004. Epub 2011 Apr 13. PMID 21489894
- [Result] Ohmaru T, Fujita Y, Sugitani M, Shimokawa M, Fukushima K, Kato K. Placental elasticity evaluation using virtual touch tissue quantification during pregnancy. Placenta. 2015 Aug;36(8):915-20. doi: 10.1016/j.placenta.2015.06.008. Epub 2015 Jun 24. PMID 26149518
- [Result] Verwoerd-Dikkeboom CM, Koning AH, Hop WC, Rousian M, Van Der Spek PJ, Exalto N, Steegers EA. Reliability of three-dimensional sonographic measurements in early pregnancy using virtual reality. Ultrasound Obstet Gynecol. 2008 Dec;32(7):910-6. doi: 10.1002/uog.5390. PMID 18792418
- See also: Hazar, H. U., & Gültekin, S. Simulation Use in Midwifery Education. Life Sciences, 14 (3), 74-83. — https://dergipark.org.tr/tr/download/article-file/756501

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT04444258/Prot_SAP_ICF_000.pdf